CLINICAL TRIAL: NCT04871061
Title: Evaluation of Pericapsular Nerve Group Block on Positioning Pain for Spinal Anesthesia in Hip Fracture Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cigli Regional Training Hospital (Other)
Responsible Party: Principal Investigator, Hakan Aygün, principle investigator, Cigli Regional Training Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PENG55
Record Dates: First submitted 2021-04-25; First posted 2021-05-04 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Pain, Acute
Keywords: hip fracture, postoperative analgesia, positioning pain
MeSH Terms: conditions — Acute Pain; Hip Fractures | interventions — Fentanyl

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Randomization of the study will be done by a doctor who will not participate in patient follow-up with closed envelopes using computer generated randomization codes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PENG Block (Active Comparator): For patients with hip fracture and having hip surgery this study evaluates the analgesic effects of Pericapsular Nerve Group (PENG) block for positioning before spinal anesthesia.
  Interventions: Procedure: PENG Block
- Control (Active Comparator): in this group, standardised opioid doses (drug: Fentanyl) will be used for analgesia for positioning pain
  Interventions: Drug: Conventional opioid analgesia (Fentanyl)

INTERVENTIONS:
Procedure: PENG Block — Pericapsular Nerve Group Block
  Arms: PENG Block
Drug: Conventional opioid analgesia (Fentanyl) — standardised intravenous opioid
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate of analgesic effects of pericapsullar nerve group block which is performed preoperatively to assist positioning patients for performance of spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* hip fracture
* aged between 35 and 90 years old

Exclusion Criteria:

* contraindications for spinal anesthesia and PENG block
* impaired cognition or dementia
* multiple fractures
* any previous analgesic administration during the last 12 hours

Ages: 35 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-05 (Actual)

PRIMARY OUTCOMES:
Pain scores on the Numeric Rating Scale (NRS) | Group A: 5 minutes after intervention (intravenous opioid), Group B: 20 minutes after intervention (PENG block)
  Changes in Numeric Rating Scale (NRS) at rest and on movement will be recorded at intervals. NRS is a unidimensional measure of pain intensity in adults. The NRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").

SECONDARY OUTCOMES:
Duration of spinal anesthesia performance | Group A: 5 minutes after intervention (intravenous opioid), Group B: 20 minutes after intervention (PENG block)
  It will be measured in "minutes", from the start of positioning maneuvers to the spinal needle removal
Quality of patient's position | Group A: 5 minutes after intervention (intravenous opioid), Group B: 20 minutes after intervention (PENG block)
  The position will be characterized as "unsatisfactory", "satisfactory", "good" or "very good"
Analgesic consumption | 24 hours
  In the postoperative period, patients will be given opioids according to their pain density with a patient-controlled device, and the daily Morphine consumption in Patient Controlled Analgesia device will be collected and compared between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Aygun, MD, Study Director — Cigli RTH
Locations (1):
- Hakan Aygün, Izmir, Turkey (Türkiye)

REFERENCES:
- [Result] Diakomi M, Papaioannou M, Mela A, Kouskouni E, Makris A. Preoperative fascia iliaca compartment block for positioning patients with hip fractures for central nervous blockade: a randomized trial. Reg Anesth Pain Med. 2014 Sep-Oct;39(5):394-8. doi: 10.1097/AAP.0000000000000133. PMID 25068412
- [Derived] Aygun H, Tulgar S, Yigit Y, Tasdemir A, Kurt C, Genc C, Bilgin S, Senoglu N, Koksal E. Effect of ultrasound-guided pericapsular nerve group (PENG) block on pain during patient positioning for central nervous blockade in hip surgery: a randomized controlled trial. BMC Anesthesiol. 2023 Sep 15;23(1):316. doi: 10.1186/s12871-023-02245-3. PMID 37715173